CLINICAL TRIAL: NCT05285332
Title: Classified Treatment Strategy for De-novo Metastatic Breast Cancer After Systemic Adjuvant Therapywhich Patients Will Benefit From Surgery
Brief Title: Classified Treatment Strategy for De-novo Metastatic Breast Cancer After Systemic Adjuvant Therapy
Acronym: CS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Yue Yu, Deputy director, Changhai Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ChanghaiHTB
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Breast Neoplasms; Treatment; Metastatic Breast Cancer; Survival
Keywords: Breast Neoplasms; de-novo metastatic breast cancer; surgical treatment
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1 Primary and metastatic lesions PCR (Experimental): surgery 1 Mastectomy OR Breast conserving surgery
  Interventions: Procedure: surgical treatment 1
- 2 Primary lesions NPCR and metastatic lesions PCR (Experimental): surgery 1 Mastectomy OR Breast conserving surgery
  Interventions: Procedure: surgical treatment 1
- 3 Primary lesions PCR and metastatic lesions NPCR (Experimental): surgery 2 Resection of metastasis
  Interventions: Procedure: surgical treatment 2
- 4 Primary lesions NPCR and metastatic lesions NPCR (Experimental): Systemic therapy Endocrine therapy or chemotherapy or targeted therapy
  Interventions: Drug: Systemic therapy

INTERVENTIONS:
Procedure: surgical treatment 1 — Mastectomy OR Breast conserving surgery
  Other Names: surgery 1
  Arms: 1 Primary and metastatic lesions PCR; 2 Primary lesions NPCR and metastatic lesions PCR
Procedure: surgical treatment 2 — Resection of metastasis
  Other Names: surgery 2
  Arms: 3 Primary lesions PCR and metastatic lesions NPCR
Drug: Systemic therapy — Endocrine therapy or chemotherapy or targeted therapy
  Arms: 4 Primary lesions NPCR and metastatic lesions NPCR

SUMMARY:
For patients with de novo stage IV breast cancer, the current debate is whether local surgery can improve the survival of patients. There is no clinical study on the classification after systemic treatment of de novo stage IV breast cancer patients. In fact, the clinical stage of tumor can change with the change of treatment. For example, the stage Ⅲ of locally advanced breast cancer can down-staging to the stage Ⅱ after systemic treatment. Similarly, patients with stage Ⅳ can down-staging to stage Ⅱ or stage Ⅲ after systemic treatment. At this time, the patient can receive surgical treatment. Therefore, this study is to first treat de novo stage IV breast cancer patients with systemic treatment, according to the response after systemic treatment to give different treatment measures（surgery or continued systemic treatment）. The investigators hope that this study will provide new ideas for the treatment of de novo stage IV breast cancer and other de novo stage IV cancers.

DETAILED DESCRIPTION:
This study analysed and summarized the outcomes of the primary and metastatic lesions after first-line systemic therapy in patients with newly diagnosed breast cancer and then inferred the timing of surgical treatment. According to the tumour heterogeneity characteristics between the primary and metastatic tumours, the investigators investigated the following A, B and C scenarios. After systemic therapy in patients with de novo metastatic breast cancer, the outcomes of primary and metastatic lesions were mainly divided into four categories (Fig. 1a, b, c, d). It is worth noting that after treatment, the four conditions of a, b, c, and d may alternate with the progression of the tumour or modification of the treatment plan. Therefore, only a proactive evaluation and timely treatment can identify the time window for tumour treatment. The time window for surgical treatment is important because, once missed, the tumour may progress with new metastatic lesions. Figure 1-a: Imaging study indicates complete remission of primary and metastatic tumours. Diagnostic surgical treatment can be performed to determine whether a pathologic complete response (PCR) is achieved and to develop a subsequent treatment plan. Figure 1-b: Imaging study indicates complete remission of the metastatic tumour with residual primary tumour. The state of the patient in this scenario could be equivalent to that of patients with early resectable breast cancer. Surgical treatment of the primary tumour should be promptly performed. Figure 1-c: Complete remission of the primary and residual metastatic tumour. Surgical treatment can be selected for isolated and resectable metastatic tumour. Figure 1-d: No remission or even progression of the primary and metastatic tumours. The systemic treatment plan should be replaced, and the surgical treatment should not be considered.

ELIGIBILITY:
Study Population Operable stage IV breast cancer patients, whose primary lesion is invasive breast cancer confirmed by pathology, and metastases can be confirmed by pathology or imaginology examination

Inclusion Criteria:

* Operable stage IV breast cancer patients,whose primary lesion is invasive breast cancer confirmed by pathology, and metastases can be confirmed by pathology or imageology examination.
* ECOG-PS 0-2.
* Bone marrow, liver and kidney should be fully functional.
* Patients didn't received the locoregional surgery of the primary tumor in de novo.
* For the patient who accepted systematic treatment before operation, the systematic treatment must be administered within a year since diagnosed.

Exclusion Criteria:

* Accompanied with other primary malignant tumors.
* More than two visceral organ involvement.
* Patients who can't plan for follow-up effectively and regularly.
* Multiple liver metastases with deranged liver function tests (SGOT/SGPT more than four times the upper normal limit).

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-05-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Overall survival (OS), which defined as the time from the beginning of diagnosis of breast cancer to the death with any causes.

SECONDARY OUTCOMES:
Distant progression free survival | 5 years
  Distant disease free survival (D-DFS), which defined as the time from the diagnosis of de novo stage IV breast cancer to the confirmed time of distant progression, or death due to any other cause.
Locoregional progression free survival | 5 years
  Defined as time between the time of diagnosis and the time of locoregional recurrence, or death occurred.

CONTACTS AND LOCATIONS:
Overall Officials: YU YUE, doctor, Study Chair — Department of thyroid and breast surgery, Changhai Hospital